CLINICAL TRIAL: NCT04865588
Title: Rotational Atherectomy Combined With Cutting Balloon to Optimize Stent Expansion in Calcified Lesions
Acronym: ROTA-CUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samin Sharma, M.D., F.A.C.C., M.S.C.A.I. (Other)
Responsible Party: Sponsor-Investigator, Samin Sharma, M.D., F.A.C.C., M.S.C.A.I., Professor of Medicine/Cardiology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 21-0532
Record Dates: First submitted 2021-04-14; First posted 2021-04-29 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: calcified plaque; angioplasty; cutting balloon
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Atherectomy, Coronary

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- rotational atherectomy + cutting balloon (Active Comparator): angioplasty with rotational atherectomy followed by cutting balloon
  Interventions: Procedure: rotational atherectomy; Device: cutting balloon
- rotational atherectomy + plain old balloon (Active Comparator): angioplasty with rotational atherectomy followed by plain old balloon
  Interventions: Procedure: rotational atherectomy; Device: plain old balloon

INTERVENTIONS:
Procedure: rotational atherectomy — angioplasty with rotational atherectomy - a rotating instrument used to break up the calcification
Device: cutting balloon — a balloon with microsurgical blades on its outer surface which make longitudinal incisions in the calcified area in order to open resistant clogs
  Arms: rotational atherectomy + cutting balloon
Device: plain old balloon — current standard treatment of stent placement
  Arms: rotational atherectomy + plain old balloon

SUMMARY:
Rotational atherectomy is an established tool to treat blocked arteries in the heart, in which the blockage is due to significant amounts of calcified material. In rotational atherectomy, a rotating instrument is used to break up the calcification before a stent is placed and helps restore blood flow to the heart. However, severely calcified regions are difficult to treat and even after treatment arteries can re-clog and major cardiac events occur. This study will test if rotational atherectomy with the addition of a cutting balloon - a balloon with microsurgical blades on its outer surface which make longitudinal incisions in the calcified area in order to open resistant clogs - will result in increased blood vessel lumen, more optimal stent expansion and decreased cardiac problems compared to current standard treatment.

DETAILED DESCRIPTION:
This is a prospective, pilot study randomizing patients with stable Coronary Artery Disease undergoing Percutaneous Coronary Intervention for a de novo calcified lesion with drug eluting stent implantation to angioplasty with rotational atherectomy followed by cutting balloon (ROTA + CBA) or rotational atherectomy followed by plain old balloon (ROTA + POBA) in a 1:1 ratio.

The clinical investigation will be conducted at 2 centers in the US. Up to 48 randomized subjects per site will be enrolled in this study. Subjects participating in this clinical investigation will be followed for 9 months. The expected duration of enrollment is approximately 6 months. The total duration of the clinical investigation is expected to be approximately 2 years.

ELIGIBILITY:
Inclusion Criteria

* Adults Patients ≥18 years of age
* Patients undergoing percutaneous coronary intervention with planned rotational atherectomy and planned drug-eluting stent implantation of a lesion with target vessel reference diameter ≥2.5 mm and ≤ 4.0mm, lesion length ≥ 5 mm and moderate to severe calcification by angiography
* Patients eligible for percutaneous coronary intervention

Exclusion Criteria

* Patients in cardiogenic shock
* Planned surgery (cardiac and non-cardiac) within 6 months after the index procedure unless the dual-antiplatelet therapy can be maintained throughout the perisurgical period
* Patients undergoing primary percutaneous coronary intervention for ST-segment elevation myocardial infarction
* Subject is pregnant, nursing, or is a woman of child-bearing potential who is not surgically sterile, < 2 years postmenopausal, or does not consistently use effective methods of contraception
* Patient has any other serious medical illness (e.g., cancer, end-stage congestive heart failure) that may reduce life expectancy to less than 12 months
* Currently participating in another investigational drug or device study
* Patients referred to coronary artery bypass grafting after heart team discussion

Angiographic Specific Exclusion Criteria:

* Lesion(s) with angulation > 45 degrees by visual estimate
* Lesion(s) stenosis through which a guidewire will not pass.
* Last remaining vessel with compromised (<30%) left ventricular function
* Saphenous vein grafts
* Angiographic evidence of thrombus
* Angiographic evidence of significant dissection at the treatment site
* Lesion(s) with previously placed stent within 10 mm (visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samin K Sharma, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - The Icahn School of Medicine at Mount Sinai, New York, New York
  - Saint Francis Hospital and Heart Center, Roslyn, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (10.0) | 72.8 (8.7) | 71.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 21 | 26 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 25 | 27 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 1 | 4
  White | 12 | 20 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Hypertension [Count of Participants; unit: Participants] | 28 | 29 | 57
Hyperlipidaemia [Count of Participants; unit: Participants] | 28 | 29 | 57
Diabetes mellitus [Count of Participants; unit: Participants] | 12 | 13 | 25
Insulin [Count of Participants; unit: Participants] | 6 | 5 | 11
Current smoker [Count of Participants; unit: Participants] | 3 | 6 | 9
Family history of coronary artery disease (CAD) [Count of Participants; unit: Participants] | 15 | 18 | 33
Peripheral arterial disease [Count of Participants; unit: Participants] | 4 | 3 | 7
Cerebrovascular disease [Count of Participants; unit: Participants] | 3 | 5 | 8
Chronic renal insufficiency [Count of Participants; unit: Participants] | 5 | 2 | 7
Left ventricular ejection fraction (LVEF) [Mean (Standard Deviation); unit: percent] | 55.6 (9.8) | 57.3 (7.6) | 56.5 (8.7)
Prior coronary artery bypass grafting (CABG) [Count of Participants; unit: Participants] | 2 | 2 | 4
Prior percutaneous coronary intervention (PCI) [Count of Participants; unit: Participants] | 20 | 20 | 40
Prior myocardial infarction (MI) [Count of Participants; unit: Participants] | 4 | 7 | 11
Prior stroke [Count of Participants; unit: Participants] | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Minimum Stent Area After Percutaneous Coronary Intervention
Description: Post-procedure minimum stent area after percutaneous coronary intervention assessed by intravascular ultrasound (IVUS)
Time Frame: Post-procedure, Day 0
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
mm^2 | 6.7 (1.7) | 6.9 (1.8)

2. Secondary Outcome: In-segment Minimum Lumen Area After Stent Implantation and Post Dilatation
Description: In-segment Minimum lumen area after stent implantation and post dilatation assessed by intravascular ultrasound
Time Frame: Post-procedure, Day 0
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
mm^2 | 5.9 (1.4) | 6.4 (1.9)

3. Secondary Outcome: Minimum Percent Stent Expansion After Percutaneous Coronary Intervention
Description: Minimum percent stent expansion after Percutaneous Coronary Intervention assessed by intravascular ultrasound
Time Frame: Post-procedure, Day 0
Measure: Mean (Standard Deviation); unit: minimum percent expansion
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
minimum percent expansion | 86.1 (17.5) | 78.6 (14.7)

4. Secondary Outcome: Mean Percent Stent Expansion After Percutaneous Coronary Intervention
Description: Mean percent stent expansion after percutaneous coronary intervention assessed by intravascular ultrasound
Time Frame: Post-procedure, Day 0
Measure: Mean (Standard Deviation); unit: mean percent expansion
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
mean percent expansion | 112.5 (19.4) | 104.2 (13.5)

5. Secondary Outcome: Number of Participants With Dissection After Percutaneous Coronary Intervention
Description: Number of Participants with Dissection after Percutaneous Coronary Intervention assessed by intravascular ultrasound.
Time Frame: Post-procedure, Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 1 | 3

6. Secondary Outcome: Number of Participants With Stent Malapposition After Percutaneous Coronary Intervention
Description: Number of Participants with Stent malapposition after Percutaneous Coronary Intervention assessed by intravascular ultrasound. Malapposition is indicated by blood visible behind stent struts. Stents may be completely or only partially malapposed depending on how much of the stent is in contact with the lumen wall.
Time Frame: Post-Procedure, Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 5 | 9

7. Secondary Outcome: Number of Participants With Dissection After Rotational Atherectomy and Cutting Balloon Angioplasty /Non-compliant Balloon Angioplasty (CBA/NCBA)
Description: Number of Participants with Dissection after Rotational atherectomy and cutting balloon angioplasty /non-compliant balloon angioplasty (CBA/NCBA) assessed by intravascular ultrasound. A dissection or tear in the vessel wall
Time Frame: Post-CBA/NCBA before stent, Day 0
Population: one participant missing imaging for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 28 | 31
Participants | 27 | 30

8. Secondary Outcome: Number of Participants With a Calcium Fracture After Rotational Atherectomy and Cutting/Plain Old Balloon
Description: Number of Participants with a Calcium fracture after Rotational atherectomy and Cutting/Plain old balloon assessed by intravascular ultrasound. A fracture within the calcified area.
Time Frame: Post-Procedure, Day 0
Population: one participant missing imaging for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 28 | 31
Participants | 14 | 7

9. Secondary Outcome: Acute Lumen Gain In-segment After Stent Implantation Assessed by Angiography
Description: Defined as the minimal luminal diameter in stent after stent implantation minus the minimal luminal diameter at baseline (prior to percutaneous coronary intervention and/or prior to stent placement).
Time Frame: Post-procedure, Day 0
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
mm | 1.0 (0.4) | 1.1 (0.3)

10. Secondary Outcome: Acute Lumen Gain In-stent After Stent Implantation Assessed by Angiography
Description: Defined as the minimal luminal diameter in segment after stent implantation minus the minimal luminal diameter at baseline (prior to percutaneous coronary intervention and/or prior to stent placement).
Time Frame: Post-procedure, Day 0
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
mm | 1.5 (0.3) | 1.6 (0.4)

11. Secondary Outcome: Percent Residual Diameter Stenosis In-segment After Stent Implantation
Description: Percent Residual diameter stenosis in-segment after stent implantation assessed by Angiography
Time Frame: Post-procedure, Day 0
Measure: Mean (Standard Deviation); unit: percent residual diameter stenosis
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
percent residual diameter stenosis | 25.8 (8.6) | 28.4 (6.8)

12. Secondary Outcome: Percent Residual Diameter Stenosis In-stent After Stent Implantation
Description: Percent Residual diameter stenosis in-stent after stent implantation assessed by Angiography
Time Frame: Post-procedure, Day 0
Measure: Mean (Standard Deviation); unit: percent residual diameter stenosis
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
percent residual diameter stenosis | 13.8 (6.5) | 14.8 (6.1)

13. Secondary Outcome: Minimum Lumen Diameter In-segment After Stent Implantation
Description: Minimum lumen diameter in-segment after stent implantation assessed by Angiography
Time Frame: Post-procedure, Day 0
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
mm | 2.1 (0.3) | 2.1 (0.4)

14. Secondary Outcome: Minimum Lumen Diameter In-stent After Stent Implantation
Description: Minimum lumen diameter in-stent after stent implantation assessed by Angiography
Time Frame: Post-procedure, Day 0
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
mm | 2.5 (0.3) | 2.5 (0.4)

15. Secondary Outcome: Number of Participants With Dissection Type B or Greater
Description: Number of Participants with Dissection Type B or greater before and after stent implantation assessed by Angiography.
Time Frame: Post-CBA/NCBA before stent and after stent, Day 0
Population: three participants missing imaging for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 28 | 29
Participants
  Post-CBA/NCBA before stent | 6 | 13
  Post-CBA/NCBA after stent | 0 | 1

16. Secondary Outcome: Number of Participants With Perforation (Ellis Type ≥2) After Stent Implantation
Description: Number of Participants with perforation (Ellis type ≥2) after stent implantation assessed by Angiography. Perforation of a vessel
Time Frame: Post-procedure, Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

17. Secondary Outcome: Number of Participants With Side Branch Closure After Stent Implantation
Description: Number of Participants with side branch closure after stent implantation assessed by Angiography. Occlusion of a side branch
Time Frame: Post-procedure, Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

18. Secondary Outcome: Number of Participants With a Balloon Rupture
Description: Device problem; Rupture of the cutting balloon or plain old balloon
Time Frame: Post-Procedure, Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

19. Secondary Outcome: Number of Participants With Blade Detachment
Description: Device problem; detachment of a blade from the cutting balloon
Time Frame: Post-Procedure, Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

20. Secondary Outcome: Number of Participants With Difficulty in Withdrawing/Advancing the Device
Description: Device problem; difficulty in moving the balloon within the vessel during the procedure
Time Frame: Post-Procedure, Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

21. Secondary Outcome: Number of Participants Who Died of All-causes (Cardiac and Non-cardiac) After Percutaneous Coronary Intervention
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

22. Secondary Outcome: Number of Participants Who Died of Cardiac Death After Percutaneous Coronary Intervention
Description: Cardiac Death
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

23. Secondary Outcome: Number of Participants Who Died of Non-Cardiac Death After Percutaneous Coronary Intervention
Description: Non-Cardiac Death
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

24. Secondary Outcome: Number of Participants With Myocardial Infarction, as Defined by the Society for Cardiovascular Angiography and Intervention (SCAI), After Percutaneous Coronary Intervention
Description: The Society for Cardiovascular Angiography and Intervention (SCAI) defines clinically relevant MI after PCI as an elevation of cardiac biomarkers (CK-MB or troponin) above specified thresholds within 48 hours of the procedure, with or without new Q waves or LBBB on ECG. This definition aims to identify meaningful ischemic injury to the myocardium that is associated with adverse clinical outcomes.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 1 | 0

25. Secondary Outcome: Percent of Participants With Myocardial Infarction, as Defined by 4th Universal Definition, After Percutaneous Coronary Intervention
Description: Myocardial infarction is defined as heart muscle damage due to lack of blood flow, based on characteristic symptoms, ECG changes, and cardiac biomarker elevation, especially troponin. Elevated levels of cardiac biomarkers, especially troponin, along with ECG changes and cardiac symptoms, indicate myocardial infarction according to the universal definition.
Time Frame: 30 days
Measure: Number; unit: percent of participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
percent of participants | 26.9 | 13.2

26. Secondary Outcome: Number of Participants With Target Lesion Revascularization After Percutaneous Coronary Intervention
Description: Revascularization
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 1 | 0

27. Secondary Outcome: Number of Participants With Target Vessel Revascularization After Percutaneous Coronary Intervention
Description: Revascularization
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 1 | 0

28. Secondary Outcome: Number of Participants With Stent Thrombosis (Definite/Probable) After Percutaneous Coronary Intervention
Description: Stent Thrombosis
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

29. Secondary Outcome: Number of Participants With Major Bleeding (BARC 3 or 5) After Percutaneous Coronary Intervention
Description: Bleeding Academic Research Consortium (BARC) Type 3
  1. Overt bleeding plus hemoglobin drop of 3 to < 5 g/dL (provided hemoglobin drop is related to bleed); transfusion with overt bleeding
  2. Overt bleeding plus hemoglobin drop < 5 g/dL (provided hemoglobin drop is related to bleed); cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring IV vasoactive agents
  3. Intracranial hemorrhage confirmed by autopsy, imaging, or lumbar puncture; intraocular bleed compromising vision
  Type 5
  1. Probable fatal bleeding
  2. Definite fatal bleeding (overt or autopsy or imaging confirmation)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

30. Secondary Outcome: Number of Participants With Vascular Complications After Percutaneous Coronary Intervention
Description: Vascular complication
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

31. Secondary Outcome: Angina Status According to Canadian Cardiovascular Society (CSS) Classification
Description: The Canadian Cardiovascular Society (CCS) grading scale is a classification system used to grade the severity of angina pectoris based on symptoms and their relationship to physical activity.
  Grade I: Ordinary physical activity like walking does not cause angina. Angina only occurs with strenuous, rapid, prolonged exertion during recreation or work.
  Grade II: Slight limitation of ordinary activity. Angina occurs when walking/climbing stairs rapidly, walking uphill, after meals, in cold/wind, under stress, or early morning. Angina occurs when walking more than 2 blocks or climbing more than 1 flight of stairs at a normal pace.
  Grade III: Marked limitation of ordinary activity. Angina occurs when walking 1-2 blocks or climbing 1 flight of stairs at a normal pace.
  Grade IV: Inability to carry out any physical activity without angina. Anginal symptoms may be present at rest.
  Higher grades indicate more limitations to activity due to angina.
Time Frame: 270 days
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: 30 days
Description: All 30 day primary outcome site-reported adverse events were collected.
Arm/Group | Rotational Atherectomy + Cutting Balloon | Rotational Atherectomy + Plain Old Balloon
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 4/29 | 4/31
Other Adverse Events (participants affected / at risk) | 24/29 | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotational Atherectomy + Cutting Balloon (N=29) | Rotational Atherectomy + Plain Old Balloon (N=31)
Myocardial Infarction (MI) (Cardiac disorders) | 1 | 2
Revascularisation (Cardiac disorders) | 1 | 0
Peri-procedural chest pain (Cardiac disorders) | 1 | 0
Staged Percutaneous Coronary Intervention (PCI) (Cardiac disorders) | 1 | 2
Kidney Stone (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotational Atherectomy + Cutting Balloon (N=29) | Rotational Atherectomy + Plain Old Balloon (N=31)
Atrial Fibrillation (Cardiac disorders) | 0 | 2
Bleeding (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Chest Pain, Not Specified (Cardiac disorders) | 1 | 1
Chromaturia (Renal and urinary disorders) | 1 | 0
Congestion (Infections and infestations) | 1 | 0
Contusion (Skin and subcutaneous tissue disorders) | 1 | 0
Diaphoresis (Endocrine disorders) | 0 | 1
Dissection Post IVUS (Injury, poisoning and procedural complications) | 1 | 0
Dissection B Post CBA/POBA (Injury, poisoning and procedural complications) | 3 | 1
Dissection B Post ROTA (Injury, poisoning and procedural complications) | 0 | 1
Dissection B Post ROTA; Dissection B Post CBA/POBA (Injury, poisoning and procedural complications) | 0 | 1
Dissection C Post CBA/POBA (Injury, poisoning and procedural complications) | 3 | 7
Dissection C Post ROTA (Injury, poisoning and procedural complications) | 0 | 1
Dissection C Post Stent (Injury, poisoning and procedural complications) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Hypertension (Cardiac disorders) | 0 | 1
Hypokalemia (General disorders) | 1 | 0
Hypotension (Cardiac disorders) | 1 | 0
Joint Swelling (General disorders) | 1 | 0
Lymphadenopathy (Immune system disorders) | 1 | 0
Myocardial Infarction (MI) (Cardiac disorders) | 2 | 2
No-Flow Post Procedure (Injury, poisoning and procedural complications) | 1 | 0
Plaque Shift (Injury, poisoning and procedural complications) | 0 | 2
Post-PCI Troponin Leak (Injury, poisoning and procedural complications) | 16 | 20
Post-PCI Troponin Leak (Staged PCI) (Injury, poisoning and procedural complications) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Slow-Flow Post CBA/POBA (Injury, poisoning and procedural complications) | 1 | 0
Slow-Flow Post ROTA (Injury, poisoning and procedural complications) | 3 | 2
Slow-Flow Post Stent (Injury, poisoning and procedural complications) | 1 | 0
Staged PCI (Cardiac disorders) | 1 | 3
Vascular Access Site Infection (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Since study is being conducted at two sites, PIs agree that study results must be published in an integrated manner reflecting results from both sites. Written consent from ISMMS is required for publication. If there is no multi-site publication within 18 months after the study has been completed or terminated at all Study locations, Pl shall have the right to publish and/or present the results of the study generated at their site.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT04865588/Prot_SAP_000.pdf